CLINICAL TRIAL: NCT06645210
Title: A Multicenter Retrospective Cohort Study on Allergic Bronchopulmonary Aspergillosis
Brief Title: Multicenter Registration Study on Allergic Bronchopulmonary Aspergillosis
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); Guangzhou Institute of Respiratory Disease (Other); Tongji Hospital (Other); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Qianfoshan Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); West China Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Xiangya Hospital of Central South University (Other); Peking Union Medical College Hospital (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Sun Yongchang, Prof, Peking University Third Hospital
Other Study IDs: M2024692
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
Keywords: cohort study
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To understand the current diagnosis and treatment status of ABPA patients, observe their clinical characteristics, prognosis, and treatment outcomes, and identify the relevant factors for poor prognosis in patients.

ELIGIBILITY:
Inclusion Criteria:

Meeting the diagnosis of ABPA according to the ABPA diagnostic criteria specified by the ISHAM-ABPA working group in 2024

Exclusion Criteria:

ABPA patients who are not first diagnosed in the center

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with ABPA
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical classification and treatment response criteria for ABPA | 1 year
  1. Acute ABPA
  2. Response
  3. Remission
  4. Treatment-dependent ABPA
  5. Advanced ABPA

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No